CLINICAL TRIAL: NCT05609838
Title: Effect Of Hot Water Foot Bath Applied İn The Early Period After Cesarean Section On Pain, Fatigue And Gas Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Oya KAPLAN, Principal Investigator, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UGaziantep-SBF-OK-01
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Cesarean Section
Keywords: Nursing; cesarean section; pain; fatigue
MeSH Terms: conditions — Pain; Fatigue

STUDY DESIGN:
Intervention Model Description: Two groups (experimental group and control group)
Who Masked: Participant
Masking Description: The researcher knew which of the participants belonged to the experimental and control groups, but the participants did not know. It is a single-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): A 15 minutes hot water foot bath was applied to the experimental group patients 3 hours after the cesarean section.Data collection tools were applied at the 5th minute, 1st hour and 2nd hour after the hot water footbath and the gas output was questioned.
  Interventions: Other: Hot water foot bath
- Control Group (No Intervention): The control group was given routine post-cesarean care without any intervention and data collection tools were applied at the same time as the experimental group.

INTERVENTIONS:
Other: Hot water foot bath — A 15 minutes hot water foot bath was applied to the experimental group patients 3 hours after the cesarean section.
  Arms: Experimental group

SUMMARY:
The aim of this research is to determine the effect of hot water foot bath applied in the early period after cesarean section on pain, fatigue and gas release.The sample of the research consisted of 80 women who gave birth by cesarean section. 'Descriptive Information Form', 'Numerical Rating Scale', 'Visual Analogue Scale for Fatigue', 'Experimental Group Patient Follow-up Form', 'Control Group Patient Follow-up Form' were used as data collection tools. It was determined that the hot water foot bath applied in the early period after cesarean section reduced the level of pain and fatigue, and had no effect on gas release.

DETAILED DESCRIPTION:
The aim of this research is to determine the effect of hot water foot bath applied in the early period after cesarean section on pain, fatigue and gas release. This research is a randomized controlled trial. The study was conducted in Gaziantep Abdulkadir Yuksel Hospital. The sample of the research consisted of 80 women who gave birth by cesarean section (experimental group: 40 and control group: 40). The women in the study were randomly assigned to the experimental and control groups before starting the application. The data were collected between 01 December 2021 and 31 June 2022. 'Descriptive Information Form', 'Numerical Rating Scale', 'Visual Analogue Scale for Fatigue', 'Experimental Group Patient Follow-up Form', 'Control Group Patient Follow-up Form' were used as data collection tools. Hot water foot bath was applied to the experimental group for 15 minutes 3 hours after the cesarean section. The control group was only followed up after cesarean section. In the comparison of the experimental and control groups, chi-square for categorical variables, and independent samples t-test for numerical variables were used. Independent samples t-test was used to compare the scale scores of the experimental and control groups. In the comparison of the scale scores that were measured at different times, the Repeated Measurements Analysis of Variance was applied and the Least Significant Difference(LSD) test, which is one of the multiple comparison tests, was used. It was found that the pain level of the women after the hot water foot bath application in the experimental group was lower than that of the control group and the measurements before the application. It was determined that the fatigue levels of the women in the experimental group after the application were lower than the control group and the measurements before the application. It was determined that the application of hot water foot bath was not effective in the period of gas release after cesarean section. As a result, it was determined that the hot water foot bath applied in the early period after cesarean section reduced the level of pain and fatigue, and had no effect on gas release. During the post-cesarean section, a hot water foot bath can be recommended in nursing care.

ELIGIBILITY:
Inclusion Criteria:

* T.C. citizen of
* over 18 years old
* No history of any medical illness
* Receiving spinal anesthesia in cesarean section
* No complications during or after cesarean section
* Those who have not had any problems during pregnancy
* No mental handicap or perception problems and no communication difficulties
* Women who do not release gas before applying a hot water foot bath

Exclusion Criteria:

* Those who have intestinal discomfort during pregnancy and before pregnancy, have undergone intestinal surgery
* Gas-releasing before hot water footbath application
* sensory loss
* Wounds and/or lesions on their feet
* Those with vascular diseases

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The numerical rating scale (NRS) | at the 3rd hour after cesarean section before hot water foot bath application
  It is a frequently preferred scale because it is thought to be easy to apply. With this scale, the patient's pain is explained with numerical values. Pain severity assessment in numerical scales is applied as a rating starting with "0" and up to "10" level. Here, "0" means no pain, "10" means unbearable pain. In this assessment scale, the patient is asked to express the level of pain he/she feels at that moment with numbers.
The numerical rating scale (NRS) | at the 5th minute after the application of hot water foot bath
  It is a frequently preferred scale because it is thought to be easy to apply. With this scale, the patient's pain is explained with numerical values. Pain severity assessment in numerical scales is applied as a rating starting with "0" and up to "10" level. Here, "0" means no pain, "10" means unbearable pain. In this assessment scale, the patient is asked to express the level of pain he/she feels at that moment with numbers.
The numerical rating scale (NRS) | at the 1st hour after the application of hot water foot bath
  It is a frequently preferred scale because it is thought to be easy to apply. With this scale, the patient's pain is explained with numerical values. Pain severity assessment in numerical scales is applied as a rating starting with "0" and up to "10" level. Here, "0" means no pain, "10" means unbearable pain. In this assessment scale, the patient is asked to express the level of pain he/she feels at that moment with numbers.
The numerical rating scale (NRS) | at the 2nd hour after the application of hot water foot bath
  It is a frequently preferred scale because it is thought to be easy to apply. With this scale, the patient's pain is explained with numerical values. Pain severity assessment in numerical scales is applied as a rating starting with "0" and up to "10" level. Here, "0" means no pain, "10" means unbearable pain. In this assessment scale, the patient is asked to express the level of pain he/she feels at that moment with numbers.

SECONDARY OUTCOMES:
'Visual Analogue Scale for Fatigue (VAS-F) | at the 3rd hour after cesarean section before hot water foot bath application
  The scale consists of 18 items relating to the subjective experience of fatigue. Each item asks respondents to place an "X," representing how they currently feel, along a visual analogue line that extends between two extremes (e.g., from "not at all tired" to "extremely tired").
'Visual Analogue Scale for Fatigue (VAS-F) | at the 5th minute after the application of hot water foot bath
  The scale consists of 18 items relating to the subjective experience of fatigue. Each item asks respondents to place an "X," representing how they currently feel, along a visual analogue line that extends between two extremes (e.g., from "not at all tired" to "extremely tired").
'Visual Analogue Scale for Fatigue (VAS-F) | at the 1st hour after the application of hot water foot bath
  The scale consists of 18 items relating to the subjective experience of fatigue. Each item asks respondents to place an "X," representing how they currently feel, along a visual analogue line that extends between two extremes (e.g., from "not at all tired" to "extremely tired").
'Visual Analogue Scale for Fatigue (VAS-F) | at the 2nd hour after the application of hot water foot bath
  The scale consists of 18 items relating to the subjective experience of fatigue. Each item asks respondents to place an "X," representing how they currently feel, along a visual analogue line that extends between two extremes (e.g., from "not at all tired" to "extremely tired").

CONTACTS AND LOCATIONS:
Overall Officials: Oya KAPLAN, PhD Student, Principal Investigator — University of Gaziantep; Simge ZEYNELOĞLU, Professor, Principal Investigator — University of Gaziantep
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No